CLINICAL TRIAL: NCT03449628
Title: L. Casei DG® (Lactobacillus Paracasei CNCMI1572) in the Treatment of Patients With Irritable Bowel Syndrome: a Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo Controlled Study.
Brief Title: L. Casei DG® in Patients With Irritable Bowel Syndrome.
Acronym: PROBE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Collaborators: 1Med (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSC-DS PROBE2-IBS/17
Record Dates: First submitted 2018-02-07; First posted 2018-02-28 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L. casei DG® (Experimental): Interventions: Lactobacillus paracasei CNCMI1572 (At least 24 billion live cells per capsule)
  1 capsule, b.i.d. for 12 weeks
  Interventions: Dietary Supplement: L.casei DG
- Placebo (Placebo Comparator): Interventions : capsules for oral use, indistinguishable from active product.
  1 capsule, b.i.d. for 12 weeks
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: L.casei DG — (At least 24 billion live cells per capsule)
  1 capsule, b.i.d. for 12 weeks
  Arms: L. casei DG®
Dietary Supplement: PLACEBO — 1 capsule, b.i.d. for 12 weeks
  Arms: Placebo

SUMMARY:
To assess the effect of L. casei DG® (Lactobacillus paracasei CNCMI1572; Enterolactis® plus) on abdominal symptoms and gut microbiota metabolism/composition in non constipated patients with IBS (Irritable Bowel Syndrome). Patients will be randomized to receive L. casei DG® capsules, b.i.d. for 12 weeks the a 4 weeks Follow Up period will follow.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and ≤ 65 years
* A positive diagnosis of non constipated IBS (i.e., IBS-D and IBS-M, both males and females), according to Rome IV criteria.
* A negative outcome of colonoscopy performed within 5 years before screening if patient is at least 50 years old, or if patient meet any of the following alarm features:

  1. Has a documented weight loss within the past 6 months; or
  2. Has nocturnal symptoms; or
  3. Has a familiar history of colon cancer; or
  4. Has blood mixed with their stool (excluding blood from hemorroids).
* Negative relevant additional screening or consultation whenever appropriate
* Ability to conform to the study protocol.

Exclusion Criteria:

* Patients with IBS-C or IBS-U according to Rome IV criteria
* Presence of any relevant organic, systemic or metabolic disease (particularly significant history of cardiac, renal, neurological, psychiatric, oncology, endocrinology, metabolic or hepatic disease), or abnormal laboratory values that will be deemed clinically significant on the basis of predefined values, (i.e..liver or kidney functional levels 2-times greater than the upper reference values)
* Ascertained intestinal organic diseases, including celiac disease, food allergies or inflammatory bowel diseases (Crohn's disease, ulcerative colitis, diverticular disease, infectious colitis, ischemic colitis, microscopic colitis).
* Previous major abdominal surgery.
* Active malignancy of any type, or history of a malignancy (patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrolment are also acceptable).
* Untreated food intolerance such as ascertained or suspected lactose intolerance, as defined by anamnestic evaluation or, if appropriate, lactose breath test.
* Use of probiotics or topical and/or systemic antibiotic therapy during the last month.
* Systematic/frequent use of contact laxatives.
* Pregnant females or females of childbearing potential in the absence of effective contraceptive methods.
* Inability to conform to protocol.
* Treatment with any investigational drug within the previous 30 days.
* Recent history or suspicion of alcohol abuse or drug addiction.
* Presence of red or white flags at the Rome IV Psychosocial Alarm Questionnaire for Functional gastrointestinal Disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who have a response in pain | 12 weeks
  Patients who record on ≥ 50% of the days a reduction of ≥ 30% from their average baseline score for their worst abdominal pain.The standard 11-point numeric rating scale (from 0=none to 10=worst possible pain) will be used to measure abdominal pain.
Proportion of patients who have a response in stool consistencies | 12 weeks
  Patients who record a stool-consistency score < 5 in the same days in which they record a reduction of ≥ 30% from their average baseline score for their worst abdominal pain .For abnormal defecation, stool frequency and form will be measured using the Bristol Stool Form Scale (BSFS).

SECONDARY OUTCOMES:
Evaluation of Pain relief | 16 weeks
  reduction of ≥ 30% from baseline in the score for the worst abdominal pain on ≥ 50% of days
Evaluation of global symptom score | 16 weeks
  Improvement in the global symptom score: a score of 0 or 1, or an improvement ≥ 2 over the baseline score, on ≥ 50% of days
Relief of IBS symptoms | 16 weeks
  Adequate relief of IBS symptoms on ≥ 50% of the past weeks (a response of "yes" on ≥50% of the weeks to the following question: "Over the past week, have you had adequate relief of your IBS symptoms?)"
IBS-SSS score questionnaire (Severity Scoring System ) | 16 weeks
  To assess the severity of symptoms related to Irritable Bowel Syndrome, assessed at baseline and at the end of treatment after 12 weeks (it is considered clinically significant a score reduction of at least 50 points). The questionnaire is composed by five questions wich generate a maximum score of 100 each using prompted visual analogue scales, leading to a total possible score of 500.
Improvement in stool consistency | 16 weeks
  stool consistency score ≤ 5 assessed with BSFS (Bristol Stool Form Scale) BSFS evaluates stool form and consistency (score from 1=dry stool to 7=liquid stoo. The ideal stool is generally 3 or 4)
Satisfaction with treatment | 16 weeks
  Overall satisfaction with treatment assessed by VAS scale (Visual Analogue Scale)
Quality of life | 16 weeks
  Quality of life assessment by validated Short-Form 12 Items Health Survey (SF-12) on a scale of 0 to 100
Intake of rescue medication | 16 weeks
  type and frequencies of rescue medication
gut microbiota composition | 16 weeks
  Evaluation of changes in the gut microbiota composition and the relative abundance of bacterial OTUs (Operational Taxonomic Unit).
Short Chain Fatty Acids (SCFA) | 16 weeks
  Evaluation of Short Chain Fatty Acids levels in fecal samples
Free Aminoacids | 16 weeks
  Evaluation of Free aminoacids levels in fecal samples
Biogenic Amines | 16 weeks
  Evaluation of biogenic amines levels in fecal samples
Gut permeability for zonulin | 16 weeks
  evaluation of serum levels of zonulin
Gut permeability for citrulline | 16 weeks
  evaluation of serum levels of citrulline
Gut permeability for PV-1 (Plasmalemma vesicle-associated) protein | 16 weeks
  evaluation of serum levels of PV-1 (Plasmalemma vesicle-associated) protein
L. casei DG® strain in the feces | 16 weeks
  the recovery of L. casei DG® strain in the feces

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Barbara, MD, Principal Investigator — AUO Sant'Orsola Malpighi Bologna (Gastroenterology)
Locations (20):
- Italy (20):
  - A.O. Bolognini, Seriate, BG
  - A.O. "G. Brotzu"- Ospedale San Michele, Cagliari, CA
  - AOU di Cagliari - Policlinico di Monserrato, Cagliari, CA
  - Ospedale Valduce, Como, CO
  - ASST-FTB-Sacco, Milan, MI
  - Policlinico San Donato, San Donato Milanese, MI
  - Ospedale Sant'Andrea, Vercelli, VC
  - Gastroenterologia Universitaria Policlinico Giovanni XXIII, Bari
  - Azienda ULSS 1, Belluno
  - Azienda Ospedaliero-Universitaria S. Orsola Malpighi, Bologna
  - Ospedale SS. Annunziata, Chieti
  - Fondazione IRCCS Policlinico, Milan
  - Policlinico, Napoli
  - Policlinico Federico II, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - U.O. Gastroenterologia Universitaria, Pisa
  - Policlinico Universitario Campus Biomedico, Roma
  - A.O. San Camillo-Forlanini, Roma
  - Ospedale Sant'Andrea, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Barbara G, Feinle-Bisset C, Ghoshal UC, Quigley EM, Santos J, Vanner S, Vergnolle N, Zoetendal EG. The Intestinal Microenvironment and Functional Gastrointestinal Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00219-5. doi: 10.1053/j.gastro.2016.02.028. Online ahead of print. PMID 27144620
- [Background] Spiller R, Garsed K. Postinfectious irritable bowel syndrome. Gastroenterology. 2009 May;136(6):1979-88. doi: 10.1053/j.gastro.2009.02.074. Epub 2009 May 7. PMID 19457422
- [Background] Schoepfer AM, Schaffer T, Seibold-Schmid B, Muller S, Seibold F. Antibodies to flagellin indicate reactivity to bacterial antigens in IBS patients. Neurogastroenterol Motil. 2008 Oct;20(10):1110-8. doi: 10.1111/j.1365-2982.2008.01166.x. Epub 2008 Aug 6. PMID 18694443
- [Background] Langhorst J, Junge A, Rueffer A, Wehkamp J, Foell D, Michalsen A, Musial F, Dobos GJ. Elevated human beta-defensin-2 levels indicate an activation of the innate immune system in patients with irritable bowel syndrome. Am J Gastroenterol. 2009 Feb;104(2):404-10. doi: 10.1038/ajg.2008.86. Epub 2009 Jan 20. PMID 19174795
- [Background] Pimentel M, Morales W, Rezaie A, Marsh E, Lembo A, Mirocha J, Leffler DA, Marsh Z, Weitsman S, Chua KS, Barlow GM, Bortey E, Forbes W, Yu A, Chang C. Development and validation of a biomarker for diarrhea-predominant irritable bowel syndrome in human subjects. PLoS One. 2015 May 13;10(5):e0126438. doi: 10.1371/journal.pone.0126438. eCollection 2015. PMID 25970536
- [Background] Rajilic-Stojanovic M, Biagi E, Heilig HG, Kajander K, Kekkonen RA, Tims S, de Vos WM. Global and deep molecular analysis of microbiota signatures in fecal samples from patients with irritable bowel syndrome. Gastroenterology. 2011 Nov;141(5):1792-801. doi: 10.1053/j.gastro.2011.07.043. Epub 2011 Aug 5. PMID 21820992
- [Background] Jalanka-Tuovinen J, Salojarvi J, Salonen A, Immonen O, Garsed K, Kelly FM, Zaitoun A, Palva A, Spiller RC, de Vos WM. Faecal microbiota composition and host-microbe cross-talk following gastroenteritis and in postinfectious irritable bowel syndrome. Gut. 2014 Nov;63(11):1737-45. doi: 10.1136/gutjnl-2013-305994. Epub 2013 Dec 5. PMID 24310267
- [Background] Simren M, Barbara G, Flint HJ, Spiegel BM, Spiller RC, Vanner S, Verdu EF, Whorwell PJ, Zoetendal EG; Rome Foundation Committee. Intestinal microbiota in functional bowel disorders: a Rome foundation report. Gut. 2013 Jan;62(1):159-76. doi: 10.1136/gutjnl-2012-302167. Epub 2012 Jun 22. PMID 22730468
- [Background] Moayyedi P, Ford AC, Talley NJ, Cremonini F, Foxx-Orenstein AE, Brandt LJ, Quigley EM. The efficacy of probiotics in the treatment of irritable bowel syndrome: a systematic review. Gut. 2010 Mar;59(3):325-32. doi: 10.1136/gut.2008.167270. Epub 2008 Dec 17. PMID 19091823